CLINICAL TRIAL: NCT02363608
Title: Caring Canines: Outcomes From an Animal Assisted Activity Program on Patients and Staff on an Inpatient Surgical Oncology Unit
Brief Title: Animal Assisted Activity Program on Patients and Staff on an Inpatient Surgical Oncology Unit
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-010
Record Dates: First submitted 2015-02-05; First posted 2015-02-16 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Care
Keywords: Canine-Assisted; 15-010; post surgery patients
MeSH Terms: interventions — BaseLine dental cement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- standard post surgery care: An initial cohort of consecutive patients admitted to the 15th floor of the hospital on a Monday or Tuesday will form the usual care control arm of the study. Once this cohort is completed, the Caring Canines program will start.
  Interventions: Other: standard post surgery care
- Caring Canines program: Once the standard of care cohort is completed, the Caring Canines program will start making visits on the 15th floor and a second cohort of consecutive patients admitted to M15 on a Monday or Tuesday will form the intervention (experimental) arm of the study.patients admitted to M15 on a Monday or Tuesday will form the intervention (experimental) arm of the study.
  Interventions: Behavioral: Caring Canine program; Behavioral: baseline and post assessment
- staff canine-assisted: For the staff portion of this study a longitudinal pre and post intervention design will be used. Baseline staff assessments will occur prior to the Caring Canine program being implemented on the unit. The assessments include questions about compassion satisfaction and compassion fatigue as well as some open ended questions about your thoughts on the Caring Canines program. Post assessment will occur after the program has been active on the unit for at least 6 weeks. Only staff who work at least one Monday - Friday day shift each week will be eligible to participate.
  Interventions: Behavioral: Caring Canine program; Behavioral: baseline and post assessment

INTERVENTIONS:
Other: standard post surgery care
  Groups: standard post surgery care
Behavioral: Caring Canine program — The therapy dogs who visit at MSKCC. A visit by a therapy dog typically lasts about 10-15 minutes with the patient interacting with the therapy dog while the dog is supervised by the handler.
  Groups: Caring Canines program; staff canine-assisted
Behavioral: baseline and post assessment — The baseline and post assessment will include the Professional Quality of Life Scale (ProQOL R-IV) (Stamm, 1997-2005) and qualitative questions.
  Groups: Caring Canines program; staff canine-assisted

SUMMARY:
The purpose of this study is to describe the effects of canine-assisted activity visits on patients and staff in a hospital setting. The Caring Canines program uses dogs who have been trained to be obedient, calm and comforting. It involves a visit by a volunteer (called the dog's handler) and the volunteer's dog that has been trained and tested to have a good personality and to follow commands. A visit typically lasts about 10-15 minutes with the patient interacting with the dog while the dog is supervised by the handler. Memorial Sloan Kettering currently has Caring Canine dogs visit patients but the investigators don't yet know the impact of these visits on patients and staff. The investigators would like to see how the Caring Canine visits impact a patients' mood, including anxiety, stress, and sense of well-being. Two groups of patients will take part in this study - the first group will receive standard post surgery care and will not receive a visit from the Caring Canines program and the second group will receive daily visits (Tuesday -Friday) from the Caring Canines program while they are on M15. The purpose of this study is to look at differences in well-being between patients who have the visits with the dogs and patients who do not.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Age greater than 21
* Admitted to M15 following a Monday or Tuesday surgery
* Ability to speak and read English.

Staff

* Age greater than 21
* Works at least one day shift a week on M15
* Ability to speak and read English

Exclusion Criteria:

Patients

* Self reported allergy to dogs
* Medical need to be in an isolation room
* Medical need to be in a Protective Environment room .

Staff

* Self reported allergy to dogs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Staff and inpatients on the 15th floor.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
change from baseline in the follow-up PHQ-4 scores | 1 year
  The PHQ-4 is an ultra-brief self-report questionnaire that consists of a 2-item depression scale and a 2 item anxiety scale. Among the control and intervention groups to assess psychological effects of the program. Responses on the pain scale will assess physiological effects, and responses on the open-ended questions will identify patient-perceived benefits of the program
difference in baseline and follow-up ProQOL scores (For Staff) | 1 year
  (Compassion Satisfaction score and Burnout score) to assess change in work satisfaction due to the program, and responses on the qualitative questions will address staff-perceived benefits of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Ginex, EdD, RN, OCN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/